CLINICAL TRIAL: NCT00859183
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Investigating the Impact of Oral Sirolimus on Restenosis Prevention in Patients With In-Stent Restenosis.
Brief Title: Oral Sirolimus for In-Stent Restenosis
Acronym: OSIRIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Albert Schömig, Deutsches Herzzentrum Muenchen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. S01101
Record Dates: First submitted 2009-03-06; First posted 2009-03-10 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Coronary Restenosis
Keywords: in-stent restenosis; stents; sirolimus
MeSH Terms: conditions — Coronary Restenosis | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): cumulative loading dose of 8 mg of sirolimus two days prior to and the day of repeat intervention followed by maintenance therapy of 2 mg/day for 7 days
  Interventions: Drug: Sirolimus
- 2 (Active Comparator): cumulative loading dose of 24 mg of oral sirolimus two days prior to and the day of repeat intervention followed by maintenance therapy of 2 mg/day for 7 days
  Interventions: Drug: Sirolimus
- 3 (Placebo Comparator): oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — cumulative loading dose of 8 mg of oral sirolimus two days prior to and the day of repeat intervention followed by maintenance therapy of 2 mg/day for 7 days
  Other Names: Rapamune
  Arms: 1
Drug: Sirolimus — cumulative loading dose of 24 mg of oral sirolimus two days prior to and the day of repeat intervention followed by maintenance therapy of 2 mg/day for 7 days
  Other Names: Rapamune
  Arms: 2
Drug: Placebo — Placebo oral
  Arms: 3

SUMMARY:
Despite recent advances in interventional cardiology including the success of drug-eluting stents in de-novo coronary lesions, the treatment of in-stent restenosis remains a challenging clinical issue. Given the efficacy of the systemic sirolimus administration to prevent neointimal hyperplasia in animal models and to halt and even reverse the progression of allograft vasculopathy, the aim of the present double-blind, placebo-controlled study was to evaluate the efficacy of a 10-day oral sirolimus treatment with two different loading regimens for the prevention of recurrent restenosis in patients with in-stent restenosis.

DETAILED DESCRIPTION:
Three-hundred symptomatic patients with in-stent restenotic lesions were randomly assigned to one of three treatment arms: placebo, usual dose or high dose sirolimus. Patients received a cumulative loading dose of 0, 8 or 24 mg of sirolimus two days prior to and the day of repeat intervention followed by maintenance therapy of 2 mg/day for 7 days. Angiographic restenosis at 6-months angiography was the primary end point of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angina pectoris or exercise-induced ischemia in the presence of angiographically significant in-stent-restenosis in native coronary arteries.

Exclusion Criteria:

* Patients with acute coronary syndromes or with severe infectious diseases the presence of severe kidney failure (serum creatinine > 2.2 mg/dl) contraindications to sirolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2001-10; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Angiographic restenosis | 6 months

SECONDARY OUTCOMES:
The combined incidence of death and myocardial infarction as well as target vessel revascularization | one year

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen; Albert Schömig, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (3):
- Germany (3):
  - Medizinische Klinik I, Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - Deutsches Herzzentrum, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Result] Hausleiter J, Kastrati A, Mehilli J, Vogeser M, Zohlnhofer D, Schuhlen H, Goos C, Pache J, Dotzer F, Pogatsa-Murray G, Dirschinger J, Heemann U, Schomig A; OSIRIS Investigators. Randomized, double-blind, placebo-controlled trial of oral sirolimus for restenosis prevention in patients with in-stent restenosis: the Oral Sirolimus to Inhibit Recurrent In-stent Stenosis (OSIRIS) trial. Circulation. 2004 Aug 17;110(7):790-5. doi: 10.1161/01.CIR.0000138935.17503.35. Epub 2004 Aug 9. PMID 15302787
- [Derived] Kufner S, Hausleiter J, Ndrepepa G, Schulz S, Bruskina O, Byrne RA, Fusaro M, Kastrati A, Schomig A, Mehilli J; OSIRIS Trial Investigators. Long-term risk of adverse outcomes and new malignancies in patients treated with oral sirolimus for prevention of restenosis. JACC Cardiovasc Interv. 2009 Nov;2(11):1142-8. doi: 10.1016/j.jcin.2009.08.015. PMID 19926058